CLINICAL TRIAL: NCT01284868
Title: An Exploratory Study Into the Mechanism of Mirabegron-induced Cardiovascular Effects in Healthy Male Subjects.
Brief Title: A Study in Healthy Young Men to Look at What Drives the Cardiovascular Effects After Dosing With Mirabegron.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Disclosure Office Europe, Astellas Pharma Europe BV
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 178-CL-053; 2006-004653-14 (EudraCT Number)
Record Dates: First submitted 2011-01-23; First posted 2011-01-27 (Estimated); Last update posted 2013-07-03 (Estimated); Status verified 2011-01

CONDITIONS: Healthy Volunteers; Pharmacodynamics of Mirabegron
Keywords: Mechanisms of Pharmacological Action; Pharmacodynamics; Pharmacokinetics
MeSH Terms: interventions — mirabegron; Bisoprolol; Propranolol

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mirabegron (Experimental)
  Interventions: Drug: mirabegron; Drug: Bisoprolol; Drug: propranolol; Drug: placebo

INTERVENTIONS:
Drug: mirabegron — oral
  Other Names: YM178
Drug: Bisoprolol — oral
Drug: propranolol — oral
Drug: placebo — oral

SUMMARY:
To explore what is driving heart-rate increases after dosing with mirabegron. Subjects will be given a beta-blocker at the same time as mirabegron.

DETAILED DESCRIPTION:
Impedance cardiography parameters will be assessed and compared when mirabegron (or placebo), is taken in combination with a selective beta-blocker, a non-selective beta-blocker or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index between 20.0 and 28.5 kg/m2, inclusive
* Subject is genotyped as an extensive metabolizer for CYP2D6
* Subject agrees to sexual abstinence and/or use of a highly effective method of birth control from screening until 3 months after last dose of study medication. Examples of effective methods:

  * subject's sexual partner has been surgically sterilized (for at least 3 months prior to screening), or
  * subject/subject's sexual partner is using standard oral contraception or is practicing two (2) of the following contraceptive methods:
  * diaphragm with spermicide
  * intrauterine device
  * condoms in combination with a spermicidal cream

Exclusion Criteria:

* Known or suspected hypersensitivity to mirabegron, propranolol or bisoprolol, or any components of the formulations used
* Any of the liver function tests (i.e. ALT, AST) above the upper limit of normal at repeated measures
* Any clinically significant history of bronchospasm, asthma, eczema, allergic rhinitis during the pollen season, any other allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever)
* Any clinically significant history of sinus bradycardia, first and second degree atrioventricular block, metabolic acidosis, Raynaud's disease, cardiogenic shock, right ventricular failure secondary to pulmonary hypertension, bronchospasms, angina, peripheral arterial occlusive disease, overt cardiac failure, congestive heart failure, sick sinus syndrome or any other cardiovascular or ECG abnormalities
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Abnormal heart rate and/or blood pressure measurements at the pre-study visit as follows: Heart rate <50 or >90 bpm; mean systolic blood pressure <90 or >140 mmHg; mean diastolic blood pressure <40 or >90 mmHg (blood pressure measurements taken in triplicate after subject has been resting in supine position for 5 minutes; heart rate will be measured automatically)
* A marked baseline prolongation of QT/QTc interval after repeated measurements of > 430 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome
* PR interval > 200 ms or < 120 ms
* Evidence of second- or third-degree atrioventricular block
* Electrocardiographic evidence of complete left bundle branch block (LBBB), right bundle branch block or incomplete LBBB
* Intraventricular conduction delay with QRS duration > 120 ms
* Pathological Q-waves (defined as Q-wave > 40 ms or depth greater than 0.4 - 0.5 mV)
* Evidence of ventricular pre-excitation
* Use of any prescribed or OTC drugs (including vitamins, natural and herbal remedies, e.g. St. John's Wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse within 3 months prior to admission to the Clinical Unit
* History of smoking more than 10 cigarettes (or equivalent amount of tobacco) per day within 3 months prior to admission to the Clinical Unit
* History of drinking more than 21 units of alcohol per week (1 unit = 200 ml of beer or 25 ml of spirits or 75 ml of wine) within 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2
* Subjects who, in the opinion of the investigator, are not likely to complete the trial for any reason
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life
* Any clinical condition, which, in the opinion of the investigator would not allow safe completion of the study

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2009-07; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Plasma renin activity | 12 hours
Impedance cardiography | 12 hours

SECONDARY OUTCOMES:
Pharmacokinetic assessment of mirabegron by analysis of plasma samples | 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- Paris, France